CLINICAL TRIAL: NCT02793921
Title: Influence of Exercise on Neurocognitive Function in Breast Cancer
Brief Title: Exercise Program in Cancer and Cognition
Acronym: EPICC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Catherine M. Bender, PhD, RN, FAAN, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY19080223; 1R01CA196762-01A1 (NIH)
Record Dates: First submitted 2016-05-20; First posted 2016-06-08 (Estimated); Results first posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer
Keywords: Alteration; Cognitive Function; Exercise
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Moderate-intensity aerobic exercise (Experimental): Participants engage in a supervised 6-month moderate-intensity aerobic exercise intervention.
  Interventions: Behavioral: Moderate-Intensity Aerobic Exercise Intervention
- Usual Care (No Intervention): Physical activity neither limited nor withheld. Participants engage in activity in the same manner as if they were not part of an active intervention.

INTERVENTIONS:
Behavioral: Moderate-Intensity Aerobic Exercise Intervention — The intervention is moderate-intensity aerobic exercise. Walking on a motorized treadmill will be the encouraged mode of exercise; however participants may use other equipment or home exercise. Participants will begin by exercising 10-15 minutes for 3 days/week during the first 2 weeks and gradually increase the duration for the following 4 weeks until they reach 40-50 minutes per session/3 days per week. This level is then maintained for the remainder of the 6 months. The rate of increase will be tailored based on baseline cardiorespiratory fitness and response to exercise. All sessions start and end with a vital sign check (in-person) and 5-10 minutes warm-up/cool-down. Trained exercise physiologists will supervise all exercise sessions and closely monitor adherence, intensity, and safety when sessions are completed in-person, or through regular communication when home-based exercise is warranted (due to COVID-19).
  Arms: Moderate-intensity aerobic exercise

SUMMARY:
This randomized control trial will examine whether a well-controlled and monitored exercise intervention improves cognitive function in postmenopausal women with early-stage breast cancer and will explore whether neuroimaging metrics of brain health, pro-inflammatory biomarkers and symptoms (fatigue, sleep problems, depression, anxiety) mediate the effects of exercise on cognitive function. Furthermore, the study will explore whether the magnitude of the improvements in cognitive function are modified by estradiol levels.

DETAILED DESCRIPTION:
The specific aims include:

1. Compared to usual care, examine whether the 6-month exercise intervention improves cognitive function in postmenopausal women with early stage breast cancer.

   Hypothesis 1. Exercise will improve cognitive function in women in a domain specific fashion such that attention, executive and memory functions will be influenced more than other domains.
2. Compared to usual care, examine the direct effects of exercise on neuroimaging metrics of brain health including regional gray matter volume, white matter architecture and functional dynamics of the brain and the pro-inflammatory biomarkers (IL-6 as primary outcomes; TNF-α as secondary), and explore the direct effects of exercise on symptoms (fatigue, sleep problems, depression, anxiety).

   Hypothesis 2. Exercise will improve neuroimaging metrics of brain health and pro-inflammatory biomarkers.
3. Compared to usual care, explore whether the effects of exercise on cognitive function are mediated by a) neuroimaging metrics of cognitive function, b) IL-6 and TNF-α levels and c) symptoms (fatigue, sleep problems, depression, anxiety), and moderated by E2 levels.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal female
2. Maximum age 80 years
3. Able to speak and read English
4. Minimum completion of 8 years of education
5. Diagnosed with Stage 0, 1, 2 or 3a Breast Cancer
6. Within 2 years post-completion of primary treatment
7. At least two weeks post-breast conserving surgery or three weeks post-breast conserving surgery with sentinel lymph node biopsy or four weeks post-mastectomy

Exclusion Criteria:

1. Prior treatment with cancer chemotherapy, central nervous system radiation, or intrathecal therapy 2. Clinical evidence of distant metastases 3. Self-report of hospitalization for psychiatric illness within the last two years 4. History of neurologic illness 5. Any of the following breast cancer surgery complications unless approved by the participant's health care provider: persistent seroma requiring aspiration, wound dehiscence, infection, prolonged drain output, lymphedema 6. Reconstructive surgery unless approved by the participant's health care provider 7. Any significant medical condition that would preclude them from exercising (e.g., uncontrolled diabetes, congestive heart failure, angina, uncontrolled arrhythmia or other symptoms that indicate increased risk for an acute cardiovascular or respiratory event) If necessary, we will verify this information with a participant's health care provider 8. Eating disorders or a history of substance abuse 10. Any use of an assisted walking device 11. Recent history of falls or balance problems

Additional Exclusion Criteria for Neuroimaging subgroup:

1. Presence of metal implants (i.e., pacemaker, some stents)

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine M Bender, PhD, Principal Investigator — University of Pittsburgh; Kirk I Erickson, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
At the completion of the intervention, after investigators have been un-blinded to group status, and after the testing and publication of the primary aims and hypotheses, the investigators will provide de-identified data to interested investigators provided that they closely consult with Drs. Bender and Erickson with respect to study design, analytical procedures, and to avoid overlapping research in analyses or manuscript preparation. The primary investigative team will be given priority in addressing scientific questions of interest with the collected data, but will work closely with any interested investigators in maximizing the data to address other questions of interest that could be answered by these data.

REFERENCES:
- [Derived] Liu S, Liu D, Bender CM, Erickson KI, Sereika SM, Shaffer JR, Weeks DE, Conley YP. DNA methylation associations with cognitive function in early-stage hormone receptor-positive breast cancer patients. Epigenomics. 2025 Sep;17(13):879-889. doi: 10.1080/17501911.2025.2542116. Epub 2025 Aug 6. PMID 40768266
- [Derived] Bender CM, Sereika SM, Gentry AL, Zhu Y, Wagner M, Cuglewski C, Duquette J, Grove G, Cummings M, Cho MG, Brufsky AM, Diego EJ, McAuliffe PF, Marsland AL, Conley YP, Erickson KI. Aerobic exercise and aromatase inhibitor-associated musculoskeletal symptoms: results of a randomized clinical trial. Support Care Cancer. 2025 Mar 4;33(3):244. doi: 10.1007/s00520-025-09257-4. PMID 40035875
- [Derived] Bender CM, Sereika SM, Gentry AL, Duquette JE, Casillo FE, Marsland A, Brufsky AM, Evans S, Gorantla VC, Grahovac TL, McAuliffe PF, Steiman JG, Zhu Y, Erickson KI. Physical activity, cardiorespiratory fitness, and cognitive function in postmenopausal women with breast cancer. Support Care Cancer. 2021 Jul;29(7):3743-3752. doi: 10.1007/s00520-020-05865-4. Epub 2020 Nov 19. PMID 33210238
- [Derived] Gentry AL, Erickson KI, Sereika SM, Casillo FE, Crisafio ME, Donahue PT, Grove GA, Marsland AL, Watt JC, Bender CM. Protocol for Exercise Program in Cancer and Cognition (EPICC): A randomized controlled trial of the effects of aerobic exercise on cognitive function in postmenopausal women with breast cancer receiving aromatase inhibitor therapy. Contemp Clin Trials. 2018 Apr;67:109-115. doi: 10.1016/j.cct.2018.02.012. Epub 2018 Mar 6. PMID 29501739

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Moderate-intensity Aerobic Exercise | Usual Care
Started | 77 | 76
Completed | 77 | 76
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Moderate-intensity Aerobic Exercise | Usual Care | Total
Number analyzed (Participants) | 77 | 76 | 153
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 45 | 43 | 88
  >=65 years | 32 | 33 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.44 (8.96) | 62.75 (7.25) | 62.09 (8.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 76 | 153
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 4 | 10
  White | 68 | 69 | 137
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 77 | 76 | 153
BMI, Customized [Mean (Standard Deviation); unit: kg/m^2] | 30.46 (7.21) | 31.14 (6.01) | 30.8 (6.7)
Disease Stage: DCIS, I, IIa, IIb, IIIa [Count of Participants; unit: Participants] — Breast cancer stages, defined by American College of Surgeons, retrieved from medical record.
  Stage 0=noninvasive Stage 1=tumor </=2cm, no lymph node spread Stage 2a=tumor</=2cm, spread to axillary lymph nodes or tumor 2-5cm, no axillary lymph node spread.
  Stage 2b=tumor 2-5cm, spread to 1-3 axillary lymph nodes or to lymph nodes near breastbone or tumor >5cm, no axillary lymph node spread Stage 3a=tumor >5 cm & spread to 1-3 axillary lymph nodes or to lymph nodes near breastbone.
  Increasing stages: >extent of cancer. Increasing stages indicate greater extent of breast cancer.
  Participants
    DCIS | 13 | 8 | 21
    Stage 1 | 44 | 54 | 98
    Stage 2a | 11 | 10 | 21
    Stage 2b | 6 | 1 | 7
    Stage 3a | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Cognitive Function
Description: Cognitive function was assessed with a battery of 14 measures. A data reduction technique, exploratory factor analysis with principal component extraction and varimax (orthogonal) rotation, was used to create summary factors. The cognitive factors identified included processing speed, attention, mental flexibility, working memory, learning and memory, verbal memory, and executive function were derived via this factor analysis. Individual measures with the highest loadings were included in each factor. All measures had factor loadings >0.400. Scores from the individual measures for each factor were normed based on healthy controls of similar age and education to yield a z-score and these were summed to yield an average z-score for each factor. Z-scores range from -4 to +4, where higher z-scores indicate better performance for each factor.
Time Frame: Baseline to 6 months
Measure: Least Squares Mean (Standard Error); unit: z-score
Arm/Group | Moderate-intensity Aerobic Exercise | Usual Care
Number analyzed (Participants) | 77 | 76
z-score
  Processing Speed | -0.05 (0.02) | 0.01 (0.02)
  Attention | 0.21 (0.04) | 0.17 (0.04)
  Mental Flexibility | -0.05 (0.03) | -0.07 (0.03)
  Working Memory | 0.28 (0.11) | 0.13 (0.12)
  Learning and Memory | 0.13 (0.06) | 0.05 (0.06)
  Verbal Memory | -0.17 (0.09) | -0.18 (0.09)
  Executive Function | -0.02 (0.03) | -0.02 (0.02)

2. Secondary Outcome: Total Brain Size
Description: High-resolution anatomical MPRAGE (1mm3 voxels, 256 slices) images will be used for volumetric analyses. The FreeSurfer pipeline using its longitudinal option will be employed to compute cortical volumes.
Time Frame: Baseline and 6 months
Population: The sample size for the total brain size analysis is smaller than the total number of participants because, imaging was planned on a subset of the overall sample, the impact of COVID precluded imaging for a time, the MRI machine was switched during the study, so it would have required some participants to use one imaging machine and another set with a second machine. Thus, the parameters of the sequences and the image quality would have been different between machines, and budget cuts.
Measure: Mean (Standard Deviation); unit: mm-cubed
Arm/Group | Moderate-intensity Aerobic Exercise | Usual Care
Number analyzed (Participants) | 17 | 16
mm-cubed
  Baseline | 1026742.118 (75232.467) | 1044057.647 (102747.151)
  6 Months | 1033171.625 (69084.048) | 1058477.167 (103402.622)

3. Secondary Outcome: Pro-inflammatory Cytokines
Description: Cytokine levels for interleukin-6 (IL-6) and tumor necrosis factor-alpha (TNF-alpha) were determined using high-sensitivity, quantitative sandwich enzyme immunoassay run according to manufacturer's directions. Greater pgs/ML indicate higher levels of both IL-6 and TNF-aplha.
Time Frame: Baseline to 6 months
Population: The number of participants analyzed for the pro-inflammatory cytokines, IL-5 and TNF-alpha is smaller than what is reported in the participant flow module because the impact of COVID precluded securing the blood samples for IL-6 and TNF-alpha for a time.
Measure: Mean (Standard Error); unit: pg/ML
Arm/Group | Moderate-intensity Aerobic Exercise | Usual Care
Number analyzed (Participants) | 58 | 55
pg/ML
  IL-6 | 0.47 (0.07) | 0.45 (0.07)
  TNF-a | 0.07 (0.01) | 0.09 (0.01)

4. Secondary Outcome: Peak VO2
Description: Fitness will be measured by submaximal VO2 test. The submaximal test is similar to the full test, but stops at 85% of the age-predicted heart rate. The protocol involves walking at a self-selected pace between 2.0-4.0 mph with increasing grade increments of 2% every two minutes. The test is terminated when the subject reaches 85% of their age-predicted heart rate or at volitional exhaustion. Higher levels (ml/kg/minute) indicate better peak VO2.
Time Frame: Baseline and 6 months
Population: The number of participants analyzed for peak VO2 is smaller than what is reported in the participant flow module because the impact of COVID precluded securing VO2 for a time.
Measure: Mean (Standard Error); unit: ml/kg/minute
Arm/Group | Moderate-intensity Aerobic Exercise | Usual Care
Number analyzed (Participants) | 62 | 66
ml/kg/minute
  Baseline | 17.31 (0.42) | 17.72 (0.48)
  6 months | 18.44 (0.38) | 19.74 (3.88)

5. Secondary Outcome: Estradiol (E2) Levels
Description: E2 was determined by a competitive binding immunoassay, according to manufacturer's directions. Greater pgs/ML indicate higher levels of estradiol.
Time Frame: Baseline to 6 months
Population: The number of participants analyzed for estradiol is smaller than what is reported in the participant flow module because the impact of COVID precluded securing blood samples for estradiol for a time.
Measure: Mean (Standard Error); unit: pg/ML
Arm/Group | Moderate-intensity Aerobic Exercise | Usual Care
Number analyzed (Participants) | 58 | 55
pg/ML | 0.48 (0.07) | 0.67 (0.12)

6. Secondary Outcome: Fatigue
Description: The Fatigue 8a Patient Reported Outcomes Measurement Information System (PROMIS) short form was used to measure fatigue. It consists of 8 items on which participants respond using a 5-point Likert scale. The scores range from 0 to 24 with higher scores indicating greater fatigue.
Time Frame: Baseline and 6 months
Population: The sample size for the analysis of the fatigue data is smaller than the total numbers in the Participant Flow module because the impact of COVID precluded securing fatigue measurement for a time.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Moderate-intensity Aerobic Exercise | Usual Care
Number analyzed (Participants) | 76 | 66
score on a scale
  Baseline | 18.60 (0.82) | 18.90 (0.86)
  6 months | 17.81 (0.92) | 16.83 (0.97)

7. Secondary Outcome: Anxiety
Description: The eight-item Anxiety 8a PROMIS short form was used to measure anxiety. Participants rate each item on a scale from 1 to 5. The score is the total of the responses with higher scores indicating greater anxiety. The range of scores is 5 to 40.
Time Frame: Baseline to 6 months
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Moderate-intensity Aerobic Exercise | Usual Care
Number analyzed (Participants) | 77 | 76
units on a scale | 1.85 (0.36) | 1.55 (0.28)

8. Secondary Outcome: Sleep Problems
Description: Sleep problems were measured using global score of the Pittsburgh Sleep Quality Index (PSQI). The PSQI is a self-report measure that consists of 19 items. Each item is weighted on a 0-3 interval scale. The PSQI global score ranges from 0 to 21, where lower scores indicate better sleep quality, and higher scores indicate poorer sleep quality.
Time Frame: Baseline to 6 months
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Moderate-intensity Aerobic Exercise | Usual Care
Number analyzed (Participants) | 77 | 76
units on a scale | 12.21 (1.57) | 13.36 (1.62)

9. Secondary Outcome: Depressive Symptoms
Description: Depressive symptoms will be measured using the Beck Depression Inventory II (BDI II). The 21-item BDI II is a self-report measure on which participants rate depressive symptoms on a four-point scale. The BDI II score ranges from 0 to 63 with higher scores indicating greater depressive symptomatology.
Time Frame: Baseline to 6 months
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Moderate-intensity Aerobic Exercise | Usual Care
Number analyzed (Participants) | 77 | 76
units on a scale | 5.51 (0.71) | 5.27 (0.61)

10. Other Pre Specified Outcome: Change in White Matter Microstructure
Time Frame: Baseline and 6 months
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Changes in Prefrontal Cortex
Time Frame: Baseline and 6 months
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Changes in Task-evoked Functional MRI Outcomes
Time Frame: Baseline and 6 months
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Changes in Resting State Network
Time Frame: Baseline and 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Moderate-intensity Aerobic Exercise | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/76
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/76
Other Adverse Events (participants affected / at risk) | 0/77 | 0/76

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-14): https://cdn.clinicaltrials.gov/large-docs/21/NCT02793921/Prot_SAP_000.pdf